CLINICAL TRIAL: NCT06880796
Title: Evaluating the Effectiveness of Mindfulness-Based Therapy for SMI Implemented in a Community Mental Health Setting
Brief Title: Mindfulness-Based Therapy for Serious Mental Illness
Acronym: MBT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2412-001; R01MH136540 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Serious Mental Illness; Schizophrenia; Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based therapy (Experimental): Mindfulness-based therapy is a type of psychotherapy that will be provided in a group format for 12 weeks.
  Interventions: Behavioral: Mindfulness-based therapy
- Treatment as Usual (Active Comparator): Treatment as usually provided including pharmacotherapy, psychotherapy, and case management as indicated.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Mindfulness-based therapy — Mindfulness-based therapy provided in a group format.
  Arms: Mindfulness-based therapy
Behavioral: Treatment as Usual (TAU) — Treatment as usually provided.
  Arms: Treatment as Usual

SUMMARY:
Serious mental illness (SMI), encompassing schizophrenia-spectrum and major mood disorders, has been estimated to affect approximately 5.4% of the U.S. adult population each year. Research shows low rates of evidence-based treatment being provided to patients with SMI. This is unfortunate, because evidence-based psychological therapies have been shown to be effective for improving outcomes in SMI. One such efficacious psychological intervention is mindfulness-based therapy (MBT), which integrates mindfulness practice with cognitive-behavioral strategies to improve illness management. Previous trials conducted in the United Kingdom have shown that MBT improves symptoms and functioning in community-based outpatients with SMI, including in routine practice settings. In the U.S., most patients with SMI receive treatment at local community mental health centers (CMHCs). However, patients in CMHCs often cannot access evidence-based therapies like MBT due to the lack of trained staff able to provide these interventions. Further, previous studies of MBT have been conducted exclusively outside the U.S. It is essential to confirm that MBT is effective when delivered for patients with SMI in the U.S., and how it can be sustainably implemented in CMHCs where this clinical population is commonly treated. Thus, the investigators propose to test the effectiveness of MBT for SMI and study its implementation in a typical CMHC setting. The investigators will randomize 160 patients with SMI (psychotic-spectrum and major mood disorders) to receive treatment as usual (TAU) vs TAU plus MBT delivered by frontline clinicians in a large, diverse CMHC. The investigators will conduct blinded assessments at baseline and at 6- (mid), 12- (post), and 24-weeks (follow-up). Consistent with an experimental therapeutics approach, the investigators will examine potential mechanisms of action (e.g., mindfulness skills), as well as collect implementation-focused quantitative and qualitative data from our community partners (patients, administrators, clinicians). If found to be effective and aided by a certified training program and the implementation data collected, MBT could be adopted as a future evidence-based practice and integrated into the routine community care of patients with SMI, thereby reducing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving treatment in a community mental health center
* Diagnosed with schizophrenia-spectrum disorder or major mood disorder based on clinical interview
* Age 18 years or older
* Ability to speak and read English

Exclusion Criteria:

* Not clinically stable enough to participate in treatment.
* Established weekly mindfulness practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 24 weeks
  The interviewer-rated Brief Psychiatric Rating Scale is a measure of psychiatric symptom severity. The total score (sum of items) will be used to assess overall severity with scores ranging from 18 to 126 and higher scores indicating greater severity.

SECONDARY OUTCOMES:
WHO Quality of Life-BREF (WHOQOL-BREF) | 24 weeks
  The WHOQOL-BREF is a 26-item self-report measure of quality of life. Items are rated on a scale from 1 to 5 with total scores ranging from 26 to 130, with higher scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be uploaded to the NIMH Data Archive.